CLINICAL TRIAL: NCT02928133
Title: Prospective Registry of Non-vitamin K Antagonist Oral Anticoagulants for ThromboEmbolic Prevention in Adult Patients With Atrial Tachyarrhythmias and Congenital Heart Disease (NOTE)
Brief Title: NOACs for Atrial Tachyarrhythmias in Congenital Heart Disease
Acronym: NOTE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: The Interuniversity Cardiology Institute of the Netherlands (Other Government)
Responsible Party: Principal Investigator, Berto J Bouma, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 036.19
Record Dates: First submitted 2015-12-21; First posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Congenital Heart Defects; Atrial Fibrillation; Ectopic Atrial Tachycardia
Keywords: Non-vitamin K antagonist oral anticoagulant (NOAC); Congenital heart disease; Atrial fibrillation; Atrial tachyarrhythmia; Thromboembolism
MeSH Terms: conditions — Heart Defects, Congenital; Atrial Fibrillation; Tachycardia, Ectopic Atrial; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Rationale: Adult patients with congenital heart disease (CHD) with atrial tachyarrhythmias need to be anticoagulated. It is not known whether non-vitamin K antagonist oral anticoagulants (NOAC) in this patient group are efficient and safe.

Aim: The purpose of the NOTE registry is to evaluate the efficacy and safety of NOACs for thromboembolic prevention in atrial tachyarrhythmias in adult patients with congenital heart disease (CHD).

Methods: In this multicenter prospective registry adult CHD patients with atrial tachyarrhythmias on NOACs (switch from VKA or new on anticoagulants) will be followed for a minimum of two years.

Primary efficacy endpoints are defined as thromboembolism, i.e. the composite of ischemic stroke, systemic and pulmonary embolism and intracardiac thrombosis, and as the composite of stroke and systemic embolism. Primary safety endpoint is defined as major bleeding according to the ISTH criteria. Secondary endpoints include each thromboembolic or bleeding event analysed separately, all-cause mortality, therapy adherence, quality of life, risk assessment of stroke and evaluation of natural history of atrial tachyarrhythmia in adult CHD patients.

Primary endpoint assessment will be performed with a per protocol analysis, and demonstrated as Kaplan Meyer estimates of event free survival and event rates per year.

DETAILED DESCRIPTION:
Rationale: Adult patients with congenital heart disease (CHD) with atrial tachyarrhythmias need to be anticoagulated. It is not known whether non-vitamin K antagonist oral anticoagulants (NOAC) in this patient group are efficient and safe.

Aim: The purpose of the NOTE registry is to evaluate the efficacy and safety of NOACs for thromboembolic prevention in atrial tachyarrhythmia's in adult patients with CHD.

Methods: In this multicenter prospective registry adult CHD patients with atrial tachyarrhythmia's on NOACs will be followed for a period of two years.

Patient population: Registry population consists of CHD patients with tachyarrhythmia's, defined as atrial fibrillation (AF) or atrial tachycardia's (AT), including atrial flutter, on NOACs. Patients with new-onset atrial tachyarrhythmia's who are eligible for NOACs, will be started directly on a NOAC. Patients on vitamin K antagonists (VKA) can be switched actively to NOACs during outpatient clinic visits, in case of agreement of both patient and physician. The switch can be initiated for various reasons, including bleeding complications on VKA, unstable INR measurements, and user friendliness. Eligibility for NOAC use is defined conform clinical practice, i.e. a patient with nonvalvular atrial tachyarrhythmia's, but without a mechanical heart valve, significantly elevated risk of bleeding, impaired renal function, or pregnancy.

Registration process: Patients will be included in the registry at start of NOAC treatment. Exclusion criteria are an expected survival of less than two years and an additional indication for anticoagulation besides atrial tachyarrhythmia's. At baseline general patient characteristics will be registered. Standard echocardiography and laboratory assessments for follow-up in adult CHD patients will be recorded during the registration period. Quality of life and therapy adherence will be assessed with questionnaires. Registry follow-up will be warranted by telephone contact or during outpatient clinic visits. At each follow-up point the occurrence of pre-defined events will be recorded. A detailed description of each variable used by the registry is provided in the protocol. Anonymized data will be collected at each investigational site and entered in a central database at the main investigational site (Academic Medical Center, Amsterdam, The Netherlands).

Quality assurance: At all investigational sites the investigators are trained to the registry protocol, case report forms and registry procedures prior to enrolling subjects. The assigned monitoring investigator at the main site, will assure regular site monitoring and auditing at all investigational sites. Source data will be verified by comparing the data to medical records and case report forms in the form of a random sample. To avoid or minimize bias, an independent clinical events committee at the main investigational site, consisting of independent physicians, assesses all primary endpoint clinical events. Intermediate evaluation will take place one year after enrollment of the last patient and consists of a verification of recorded data, assessment of accuracy of patient follow-up and primary endpoint analysis.

Drop-outs: Patients who quite NOACs or are lost to follow-up are considered drop-outs. Those who (temporarily) quite NOACs will be followed until the total follow-up of 2 years will be completed. The events that occur in the period off-NOAC will not be included in the analyses. A clear description of the reason of NOAC arrest or interruption and possible alternative anticoagulant therapy is assessed.

Endpoints: Primary efficacy endpoints are defined as thromboembolism, i.e. the composite of ischemic stroke, systemic and pulmonary embolism and intracardiac thrombosis, and as the composite of stroke and systemic embolism. Primary safety endpoint is defined as major bleeding according to the ISTH criteria. Secondary endpoints include each thromboembolic or bleeding event analyzed separately, all-cause mortality, therapy adherence, quality of life, risk assessment of stroke and evaluation of natural history of atrial tachyarrhythmia in adult CHD patients.

Sample size: By using estimates of event rates in the described patient population (thromboembolism event rate of 1.4% per year, mainly on VKA; unpublished data) and a relative risk reduction of 0.81 for stroke or systemic embolism on NOACs compared to VKA [Ruff et al, Lancet 2013], a sample size of 300 patients followed for two years is necessary to demonstrate the safety of NOACs for thromboembolic prevention with a safety margin of 2.7% thromboembolic events per year.

Statistical analysis: Endpoint assessment will be performed with a per protocol analysis, and demonstrated as Kaplan Meyer (KM) estimates of event free survival and event rates per year. The results will be compared with KM estimates and event rates from a historical similar cohort on VKA in a non-inferiority assay. Drop-outs (see below) will be censored at time of drop-out in time-to-event analyses, and included for event-rate analyses up to time of drop-out. No adjustment or imputation of missing data will be performed and all available data will be presented.

ELIGIBILITY:
Inclusion Criteria:

* Atrial tachyarrhythmia
* Congenital heart disease
* Treatment with NOAC

Exclusion Criteria:

* expected survival of less than two years
* additional indication for anticoagulation besides atrial tachyarrhythmia's

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Registry population consists of CHD patients with tachyarrhythmia's, defined as atrial fibrillation (AF) or atrial tachycardia's (AT), including atrial flutter, on NOACs. Patients with new-onset atrial tachyarrhythmia's who are eligible for NOACs, will be started directly on a NOAC. Patients on vitamin K antagonists (VKA) can be switched actively to NOACs during outpatient clinic visits, in case of agreement of both patient and physician. The switch can be initiated for various reasons, including bleeding complications on VKA, unstable INR measurements, and user friendliness. Eligibility for NOAC use is defined conform clinical practice, i.e. a patient with nonvalvular atrial tachyarrhythmia's, but without a mechanical heart valve, significantly elevated risk of bleeding, impaired renal function, or pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Thromboembolism | 2 years after enrolment
  The composite of ischemic stroke, systemic and pulmonary embolism and intracardiac thrombosis
Stroke | 2 years after enrolment
Major bleeding | 2 years after enrolment
  The composite of fatal bleeding, symptomatic bleeding in a critical organ (e.g. central nervous system, retroperitoneal, pericardial, intramuscular with compartment syndrome), and bleeding of any kind with the need for >1 packed cell, or a decrease in hemoglobin of more than 2 g/l / 1,24 mmol/l. [International Society of Thrombosis and Hemostasis (ISTH) criteria]
Systemic embolism | 2 years after enrolment

SECONDARY OUTCOMES:
All-cause mortality | 2 years after enrolment
Myocardial infarction | 2 years after enrolment
  Defined as the detection of a significant rise/fall of cardiac biomarkers in association with symptoms of ischemia, ECG changes, proof of ischemia on imaging or intracoronary thrombus at angiography. [Third definition of myocardial infarction; European Society of Cardiology (ESC) 2012]
Cardiac or non-cardiac surgical and percutaneous interventions | 2 years after enrolment
Minor bleedings | 2 years after enrolment
  Defined as all bleedings that do not meet the criteria for major bleedings [ISTH criteria]
General quality of life | 2 years after enrolment
  Quality of life assessed with questionnaire SF-36
Quality of life under anticoagulation | 2 years after enrolment
  Quality of life assessed with questionnaire PACT-Q
Therapy adherence | 2 years after enrolment
  Therapy adherence assessed with questionnaire Morisky-8

OTHER OUTCOMES:
Natural history of atrial tachyarrhythmias in CHD | 2 years after enrolment
  Progression of symptoms in EHRA classification
Natural history of atrial tachyarrhythmias in CHD | 2 years after enrolment
  Change of antiarrhythmic medication
Natural history of atrial tachyarrhythmias in CHD | 2 years after enrolment
  Occurence of ablations
Natural history of atrial tachyarrhythmias in CHD | 2 years after enrolment
  Occurence of electrical cardioversion
Natural history of atrial tachyarrhythmias in CHD | 2 years after enrolment
  Occurence of heart failure described with NYHA classification
Natural history of atrial tachyarrhythmias in CHD | 2 years after enrolment
  Occurence of heart failure described by echocardiography, ejection fraction
Natural history of atrial tachyarrhythmias in CHD | 2 years after enrolment
  Occurence of heart failure by measuring NT-proBNP

CONTACTS AND LOCATIONS:
Overall Officials: Hayang Yang, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Barbara Mulder, MD PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Berto Bouma, MD PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands